CLINICAL TRIAL: NCT04222140
Title: Early Regenerative Intervention for Post-Traumatic Osteoarthritis
Acronym: ERIPTO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Affinity Health Research Institute (Other)
Collaborators: Genesis Orthopedics and Sports Medicine (Unknown); The Center for Primary Care and Sports Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERIPTO
Record Dates: First submitted 2020-01-03; First posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Post-Traumatic Osteoarthritis of Knee
Keywords: sports medicine; regenerative medicine; bone marrow derived mesenchymal stem cells; platelet rich plasma; hyaluronic acid; post-traumatic osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ERIPTO Protocol (Experimental): Protocol arm actively being studied
  Interventions: Combination Product: ERIPTO Protocol
- BMAC only (Active Comparator): bone marrow aspirate concentrate only arm
  Interventions: Biological: BMAC Only

INTERVENTIONS:
Combination Product: ERIPTO Protocol — combination biologic treatment
  Arms: ERIPTO Protocol
Biological: BMAC Only — BMAC treatment only
  Arms: BMAC only

SUMMARY:
The goal of the proposed research is to compare the ERIPTO protocol for post-traumatic osteoarthritis of the knee with that of bone marrow aspirate concentrate (BMAC) only. The investigators will also conduct a statistical regression analysis looking into factors such as time frame from initial injury, the type of injury, gender, and age when injury first occurred. The investigators plan on evaluating clinically and radiographically the effects of the ERIPTO Protocol. There will be two arms of this study. The first arm will be our protocol arm and the second arm will be our BMAC treatment only arm. The investigators plan on collecting objective data on osteoarthritis (OA) severity by taking plain films and assessing the Kellgren-Lawrence (KL) grading scheme in assessing OA severity. The investigators will also administer MRI evaluations for cartilage and meniscal growth prior to treatment and after 1 year. The investigators also plan on collecting subjective symptom scores in the form of knee injury and osteoarthritis outcomes scores (KOOS), visual analog scores (VAS), and international knee documentation criteria (IKDC) score for OA severity. The investigators plan to track changes in both subjective and objective measures of knee OA in our patients through the course of one year.

DETAILED DESCRIPTION:
The field of regenerative medicine and orthobiologics have raised the interests of many clinicians and members of the scientific community. Over the last 20 years there has been a great interest and growth in this field, a Scopus search for musculoskeletal and stem cells resulted in over 3000 documents, with more than a third being reviews. A PubMed search in the past 6 years resulted in 52 publications in the last 5 years.

Unfortunately, the fragmentation of regenerative medicine has occured with many clinicians using generalized protocols resulting in little significant clinical improvement or short-term benefits that often fade over time.

There is still a great deal of research which needs to be done to elucidate how best to utilize the various components of regenerative medicine as well as the pathophysiology of osteoarthritis.

The ERIPTO study seeks to study a proposed protocol utilizing various components of regenerative medicine including platelet rich plasma (PRP), hyaluronic acid (HA), and human bone marrow aspirate concentrate (BMAC).

In trauma and normal wound healing collagen is often the initial activator of platelets with development of platelet monolayers over the exposed collagen surfaces as seen in post-traumatic joints. This is opposed to immediate proteolytic cleavage of platelets by thrombin with subsequent immediate release of stored growth factors. Investigations of gene expression within joints following mechanical injury to articular cartilage have been studied. In a shear versus impaction model investigators found an increase in the expression of collagen type 1 following trauma to the articular surface. This expression of collagen may act as an anchor for percutaneously injected PRP in post-traumatic joints to help facilitate steady secretion of growth factors.

It is known that the average life span of a mesangial cell once delivered into a joint is around 30 days. Only 26% of transplanted cells survive within the joint. This time frame is contingent on providing a proper and hospitable environment for the cell to be injected into. In consideration of the catabolic micro-environment of osteoarthritis it is evident that an arthritic joint, many times, harbors a molecular milieu that is not suitable or beneficial to transplanted mesangial cells and native cells including chondrocytes, type 2 collagen, the extracellular matrix, synovium, as well as subchondral progenitor cells. It can also promote osteogenic differentiation of native cartilage and lead to the progression to end stage joint disease.

Research is also coming to light regarding the inflammatory niche present in the environment at the time mesangial cells are transplanted and can hold a bearing in regards to trophic factors secreted by the mesenchymal stem cells (MSCs) as well as the immunomodulatory effects they possess. Toll like receptor stimulation on MSC polarization plays an important role in the development of a pro-inflammatory or anti-inflammatory MSC. Pro-inflammatory factors present in the milieu such as interferon (IFN) gamma or IFN alpha can influence the differentiation down the pro-inflammatory lineage of the MSC and help promote subsequent immune modulation to promote differentiation of the M1 (pro-inflammatory) macrophage, activation of CD8 T cells, as well as increased expression of pro-inflammatory chemokines such as CCL2, CXCL-9, and CXCL-10. [17] If a low level of iNOS is present that can subsequently lead to T cell activation and proliferation via cytokine-induced chemokines. Although this is largely true, expression of MSC induced IL-6 helped promote the differentiation to M2 (anti-inflammatory) lineage.

Recent research has shed light upon a novel concept within post-traumatic and arthritic joints. This is the effect the inflammatory environment and reactive oxygen species can have on native tissue dysfunction, particularly growth factors such as the TGF-B superfamily along with BMP. In 2019 investigators researched native MSC dysfunction with dysfunctional TGF-B possibly as a result of the catabolic milieu in osteoarthritis. TGF-B-induced protein (TGF-Bi) has been seen as a growth factor expressed in MSCs native to joints as well as bone marrow. It has been found to play two roles in normal chondrogenic differentiation.

In one role it stimulates proliferation and differentiation while in another role it inhibits mineralization and chondrocyte terminal differentiation. It is postulated that TGF-Bi in BM-MSCs helps regulate condensation of BM-MSCs in the early phase of chondrogenesis by bridging action between cells, collagens, and proteoglycans. In their study the investigators came to the conclusion this was achieved by modulation of adhesion molecules ITGB1, ITGB5, and NCAD. In their study the investigators were able to demonstrate the counterintuitive upregulation of TGF-Bi within the bone and articular cartilage of joints afflicted with OA, giving rise to the question of deregulation of native growth factors.

The investigators postulated either this could be the result of TGF-Bi attempting to reverse calcific changes occurring in chondrocytes of severely arthritic regions of the knee and noted an increased concentration of such within osteophytes and areas of extensive damage. The investigators also suggested a dysregulation of TGF-B family of genes within OA and did note the regulatory role TGF-Bi plays on collagen X, a marker of chondrocyte hypertrophy. Evidence is also coming to light of multiple MSC niches which exist within joints that assist in maintaining cartilage integrity and helping heal microdefects within damaged cartilage. The investigators noted among the MSCs, TGF-Bi was down regulated within the infrapatellar fat pad and BM-MSCs from OA joints and noted that whether BM-MSCs efficiency to repair cartilage lesions in vivo warrants further investigation.

The role of reactive oxygen species play in dysregulation of native BMP within musculoskeletal conditions has also been studied. The investigators discussed how low levels of ROS are required to maintain undifferentiated MSCs and how ROS (generated by NOX-2 and NOX-4) and BMP play crucial physiological roles in chondrogenesis. In a discussion regarding osteonecrosis and osteoarthritis the investigators note necrotic lesions lead to the increased production of free oxygen radical (O-, H202) with subsequent increased production of BMP-2, seen in necrotic lesions and damaged cartilage from OA patients. Increased H2O2 levels, produced by either NOX activation or inflammation, induce NF-kB activation which enhances expression of BMP-2. BMP2 stimulates proteoglycan synthesis, induces vascularization, promotes endochondral osteogenesis and has anabolic effects on chondrocyte metabolism and function, and is considered a marker for OA severity. Dysregulation of this system can lead to oxidative stress and cell dysfunction which may contribute to various pathologies.

Also, when considering MSCs capability to promote neocartilage formation, inflammation certainly plays a factor regarding its efficacy. Inflammatory factors such as TNF-alpha, IL-1B, and IL-6 hinder MSCs capability in promoting chondrogenesis by the production of excessive free radicals. The role of IL-1B in contributing to an inflammatory microenvironment has also been evaluated. These include cartilage degradation, induction of Ik-B alpha phosphorylation and subsequent nuclear translocation of nuclear factor - kappa B (NF-kB), increased reactive oxygen species (ROS) production (may also activate NF-kB), increased expression of ADAMTS-4 (inhibits gene expression of aggrecan and COMP) and reduced gene expression of anti-oxidant enzymes. The investigators discussed how elevated oxidative stress produced by these inflammatory cytokines inhibits the synthesis of cartilage matrix macromolecules (i.e. type 2 collagen and aggrecan), promotes the degradation of articular cartilage in arthritic joints, and inhibits native and implanted mesenchymal stem cell chondrogenesis.

It is now known that PRP has various influences on MSCs when combined with MSC treatment including increased proliferation rate of chondrocytes, helping promote chondrogenic differentiation, RUN X 2 inhibition, trapping of NF-KB, and affecting an overall anabolic change in the microenvironment.

It is now known that mesangial cells play an orchestrating role via paracrine related mechanisms in the expression of anabolic factors including expression of type 2 collagen, well documented anti-inflammatory and immunomodulatory role, as well as studies demonstrating recruitment of native progenitor cells versus direct differentiation. This is at the heart of what transplanted MSCs do to help in the healing process. As previously mentioned, there is only a 26% survival rate for transplanted cells and there is significant push to find bio-engineering modalities to help support the survival of transplanted MSCs. Among the modalities include transplantation of MSCs with Hyaluronan derived matrices.

Both CD44 and CD168 are involved in the regulation of growth factor signaling. Implanting MSC within an HA scaffold can help augment communication of MSCs within the joint microenvironment. The investigators also discuss the well documented pleiotropic effects of HA including anti-apoptotic, anti-inflammatory, immunosuppressive, anti-fibrotic, and chondroprotective effects. As mentioned above, with endogenous MSC dysfunction due to the presence of an inflammatory niche within osteoarthritic joints, there is an immunological response which also contributes to the arthritic milieu within joints. HA has demonstrated immunosuppressive qualities and have seen the decrease in the levels of activated T cells. There is also benefit in utilizing commercially available HA in helping normalize endogenous HA synthesis.

With the proposed ERIPTO protocol there is a logical approach to achieve more longer lasting and clinically relevant results.

ELIGIBILITY:
Inclusion Criteria:

* age 25-60 men and women
* evidence of OA both clinically and on plain films, at least KL grade 1
* no previous intra-articular treatment in the past 3 months
* In good health and active individuals exercising 1-2 times per week
* BMI 25-30
* History of meniscal, ligamentous, capsular, or articular cartilage lesions in the past
* History of impaction injury, femoral condyle fracture, tibial plateau fracture, or any OCD lesions within ≤ 5 years

Exclusion Criteria:

* Patients receiving regenerative therapies within the last 12 months
* Patients receiving corticosteroid injections within the last 3 months
* Patients with artificial joints
* Patients with secondary OA from non-traumatic mechanisms (i.e. RA or any inflammatory arthropathies)
* Patients with multiple co-morbidities that may affect the inflammatory state
* History of sleep disorders
* History of residual irregularity of articular surfaces, excessive joint instability
* History of impaction injury, femoral condyle fracture, tibial plateau fracture, or OCD lesions > 5 years
* History of malignancy, blood dyscrasias, or platelet dysfunction
* Active systemic or local infections, particularly with Klebsiella Pneumoniae, Enterococcus, and Pseudomonas

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic Changes | 1 year
  Magnetic resonance imaging evaluations pre-treatment and post-treatment measuring evidence of changes in post-traumatic osteoarthritis of the knee including articular cartilage quality, presence of subchondral bone marrow edema, presence of osteophytes, medial and lateral meniscal quality, ligamentous integrity, and presence of effusion.
Radiographic Changes | 1 year
  Kellgren Lawrence grading system will be utilized analyzing pre-treatment and post-treatment radiographs of the knee. Grading is from I-IV with I being minimal to mild disease and IV being end stage joint disease.

SECONDARY OUTCOMES:
Subjective Knee Symptom Changes | 1 year
  Three separate questionnaires will be administered at 2, 4, 6, and 12 months with the 12 month visit marking the end of the study.
  Knee Injury and Osteoarthritis Outcome Score: Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms.
Subjective Knee Symptom Changes | 1 year
  The International Knee Documentation Committee Subjective Knee Form: Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
Subjective Knee Symptom Changes | 1 year
  Visual Analogue Score: It is measured from 0 to 10 with 0 representing no pain and 10 representing severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed M Qureshi, DO, CAQSM, MRO, Principal Investigator — Affinity Health
Locations (3):
- United States (3):
  - The Center for Primary Care and Sports Medicine, Aurora, Illinois
  - Affinity Health Research Institute, Oak Brook, Illinois
  - Genesis Orthopedics and Sports Medicine, Oak Brook, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abate, Michele, Isabel Andia and Vincenzo Salini (July 1st, 2015). The Conservative Management of Osteoarthritis - Hyaluronic Acid, Platelet Rich Plasma or the Combination?, Osteoarthritis - Progress in Basic Research and Treatment, Qian Chen, IntechOpen, DOI: 10.5772/60538
- [Background] Anderson DD, Chubinskaya S, Guilak F, Martin JA, Oegema TR, Olson SA, Buckwalter JA. Post-traumatic osteoarthritis: improved understanding and opportunities for early intervention. J Orthop Res. 2011 Jun;29(6):802-9. doi: 10.1002/jor.21359. Epub 2011 Feb 11. PMID 21520254
- [Background] Andia I, Abate M. Knee osteoarthritis: hyaluronic acid, platelet-rich plasma or both in association? Expert Opin Biol Ther. 2014 May;14(5):635-49. doi: 10.1517/14712598.2014.889677. Epub 2014 Feb 17. PMID 24533435
- [Background] Angele P, Johnstone B, Kujat R, Zellner J, Nerlich M, Goldberg V, Yoo J. Stem cell based tissue engineering for meniscus repair. J Biomed Mater Res A. 2008 May;85(2):445-55. doi: 10.1002/jbm.a.31480. PMID 17729255
- [Background] Anitua E, Sanchez M, De la Fuente M, Zalduendo MM, Orive G. Plasma rich in growth factors (PRGF-Endoret) stimulates tendon and synovial fibroblasts migration and improves the biological properties of hyaluronic acid. Knee Surg Sports Traumatol Arthrosc. 2012 Sep;20(9):1657-65. doi: 10.1007/s00167-011-1697-4. Epub 2011 Oct 11. PMID 21987365
- [Background] Bain BJ. Bone marrow biopsy morbidity: review of 2003. J Clin Pathol. 2005 Apr;58(4):406-8. doi: 10.1136/jcp.2004.022178. PMID 15790706
- [Background] Barry FP, Murphy JM. Mesenchymal stem cells: clinical applications and biological characterization. Int J Biochem Cell Biol. 2004 Apr;36(4):568-84. doi: 10.1016/j.biocel.2003.11.001. PMID 15010324
- [Background] Bielecki TM, Gazdzik TS, Arendt J, Szczepanski T, Krol W, Wielkoszynski T. Antibacterial effect of autologous platelet gel enriched with growth factors and other active substances: an in vitro study. J Bone Joint Surg Br. 2007 Mar;89(3):417-20. doi: 10.1302/0301-620X.89B3.18491. PMID 17356164
- [Background] Buckwalter JA, Brown TD. Joint injury, repair, and remodeling: roles in post-traumatic osteoarthritis. Clin Orthop Relat Res. 2004 Jun;(423):7-16. PMID 15232420
- [Background] Bui, K., Duong, T., Nguyen, N., Nguyen, T., Le, V., Mai, V., Phan, N., Le, D., Phan, N., & Pham, P. (2014). Symptomatic knee osteoarthritis treatment using autologous adipose derived stem cells and platelet rich plasma: a clinical study. Biomedical Research And Therapy, 1(1):2-8.
- [Background] Chen WH, Lo WC, Hsu WC, Wei HJ, Liu HY, Lee CH, Tina Chen SY, Shieh YH, Williams DF, Deng WP. Synergistic anabolic actions of hyaluronic acid and platelet-rich plasma on cartilage regeneration in osteoarthritis therapy. Biomaterials. 2014 Dec;35(36):9599-607. doi: 10.1016/j.biomaterials.2014.07.058. Epub 2014 Aug 28. PMID 25176059
- [Background] Deakon, Timothy. "Hyaluronic Acid in the Knee: History, Characteristics and Efficacy." The Medical Xchange , 2014, pp. 7-12
- [Background] Degen RM, Bernard JA, Oliver KS, Dines JS. Commercial Separation Systems Designed for Preparation of Platelet-Rich Plasma Yield Differences in Cellular Composition. HSS J. 2017 Feb;13(1):75-80. doi: 10.1007/s11420-016-9519-3. Epub 2016 Aug 19. PMID 28167878
- [Background] Doorn J, Moll G, Le Blanc K, van Blitterswijk C, de Boer J. Therapeutic applications of mesenchymal stromal cells: paracrine effects and potential improvements. Tissue Eng Part B Rev. 2012 Apr;18(2):101-15. doi: 10.1089/ten.TEB.2011.0488. Epub 2011 Dec 22. PMID 21995703
- [Background] Everts PA, Malanga GA, Paul RV, Rothenberg JB, Stephens N, Mautner KR. Assessing clinical implications and perspectives of the pathophysiological effects of erythrocytes and plasma free hemoglobin in autologous biologics for use in musculoskeletal regenerative medicine therapies. A review. Regen Ther. 2019 May 10;11:56-64. doi: 10.1016/j.reth.2019.03.009. eCollection 2019 Dec. PMID 31193111
- [Background] Filardo G, Kon E, Roffi A, Di Matteo B, Merli ML, Marcacci M. Platelet-rich plasma: why intra-articular? A systematic review of preclinical studies and clinical evidence on PRP for joint degeneration. Knee Surg Sports Traumatol Arthrosc. 2015 Sep;23(9):2459-74. doi: 10.1007/s00167-013-2743-1. Epub 2013 Nov 26. PMID 24275957
- [Background] Glenn JD, Whartenby KA. Mesenchymal stem cells: Emerging mechanisms of immunomodulation and therapy. World J Stem Cells. 2014 Nov 26;6(5):526-39. doi: 10.4252/wjsc.v6.i5.526. PMID 25426250
- [Background] Gobbi A, Karnatzikos G, Scotti C, Mahajan V, Mazzucco L, Grigolo B. One-Step Cartilage Repair with Bone Marrow Aspirate Concentrated Cells and Collagen Matrix in Full-Thickness Knee Cartilage Lesions: Results at 2-Year Follow-up. Cartilage. 2011 Jul;2(3):286-99. doi: 10.1177/1947603510392023. PMID 26069587
- [Background] Gobbi A, Whyte GP. One-Stage Cartilage Repair Using a Hyaluronic Acid-Based Scaffold With Activated Bone Marrow-Derived Mesenchymal Stem Cells Compared With Microfracture: Five-Year Follow-up. Am J Sports Med. 2016 Nov;44(11):2846-2854. doi: 10.1177/0363546516656179. Epub 2016 Jul 29. PMID 27474386
- [Background] Goldring MB, Otero M, Plumb DA, Dragomir C, Favero M, El Hachem K, Hashimoto K, Roach HI, Olivotto E, Borzi RM, Marcu KB. Roles of inflammatory and anabolic cytokines in cartilage metabolism: signals and multiple effectors converge upon MMP-13 regulation in osteoarthritis. Eur Cell Mater. 2011 Feb 24;21:202-20. doi: 10.22203/ecm.v021a16. PMID 21351054
- [Background] Grassel S, Ahmed N. Influence of cellular microenvironment and paracrine signals on chondrogenic differentiation. Front Biosci. 2007 Sep 1;12:4946-56. doi: 10.2741/2440. PMID 17569622
- [Background] Green JD, Tollemar V, Dougherty M, Yan Z, Yin L, Ye J, Collier Z, Mohammed MK, Haydon RC, Luu HH, Kang R, Lee MJ, Ho SH, He TC, Shi LL, Athiviraham A. Multifaceted signaling regulators of chondrogenesis: Implications in cartilage regeneration and tissue engineering. Genes Dis. 2015 Dec;2(4):307-327. doi: 10.1016/j.gendis.2015.09.003. Epub 2015 Nov 6. PMID 26835506
- [Background] Greene MA, Loeser RF. Aging-related inflammation in osteoarthritis. Osteoarthritis Cartilage. 2015 Nov;23(11):1966-71. doi: 10.1016/j.joca.2015.01.008. PMID 26521742
- [Background] Grogan SP, D'Lima DD. Joint aging and chondrocyte cell death. Int J Clin Rheumtol. 2010 Apr;5(2):199-214. doi: 10.2217/ijr.10.3. PMID 20671988
- [Background] Harrell CR, Markovic BS, Fellabaum C, Arsenijevic A, Volarevic V. Mesenchymal stem cell-based therapy of osteoarthritis: Current knowledge and future perspectives. Biomed Pharmacother. 2019 Jan;109:2318-2326. doi: 10.1016/j.biopha.2018.11.099. Epub 2018 Nov 29. PMID 30551490
- [Background] Harrison S, Vavken P, Kevy S, Jacobson M, Zurakowski D, Murray MM. Platelet activation by collagen provides sustained release of anabolic cytokines. Am J Sports Med. 2011 Apr;39(4):729-34. doi: 10.1177/0363546511401576. Epub 2011 Mar 11. PMID 21398575
- [Background] Hofer HR, Tuan RS. Secreted trophic factors of mesenchymal stem cells support neurovascular and musculoskeletal therapies. Stem Cell Res Ther. 2016 Sep 9;7(1):131. doi: 10.1186/s13287-016-0394-0. PMID 27612948
- [Background] Bahrampour Juybari K, Kamarul T, Najafi M, Jafari D, Sharifi AM. Restoring the IL-1beta/NF-kappaB-induced impaired chondrogenesis by diallyl disulfide in human adipose-derived mesenchymal stem cells via attenuation of reactive oxygen species and elevation of antioxidant enzymes. Cell Tissue Res. 2018 Aug;373(2):407-419. doi: 10.1007/s00441-018-2825-y. Epub 2018 Mar 26. PMID 29582166
- [Background] Lamo-Espinosa JM, Mora G, Blanco JF, Granero-Molto F, Nunez-Cordoba JM, Sanchez-Echenique C, Bondia JM, Aquerreta JD, Andreu EJ, Ornilla E, Villaron EM, Valenti-Azcarate A, Sanchez-Guijo F, Del Canizo MC, Valenti-Nin JR, Prosper F. Intra-articular injection of two different doses of autologous bone marrow mesenchymal stem cells versus hyaluronic acid in the treatment of knee osteoarthritis: multicenter randomized controlled clinical trial (phase I/II). J Transl Med. 2016 Aug 26;14(1):246. doi: 10.1186/s12967-016-0998-2. PMID 27565858
- [Background] Lana, Jose F. Lecture Notes in Bioengineering: Platelet-Rich Plasma, Regenerative Medicine: Sports Medicine, Orthopedic, and Recovery of Musculoskeletal Injuries. Vol. 1, Springer-Verlag Berlin Heidelberg, 2014.
- [Background] Lana JF, Weglein A, Sampson SE, Vicente EF, Huber SC, Souza CV, Ambach MA, Vincent H, Urban-Paffaro A, Onodera CM, Annichino-Bizzacchi JM, Santana MH, Belangero WD. Randomized controlled trial comparing hyaluronic acid, platelet-rich plasma and the combination of both in the treatment of mild and moderate osteoarthritis of the knee. J Stem Cells Regen Med. 2016 Nov 29;12(2):69-78. doi: 10.46582/jsrm.1202011. eCollection 2016. PMID 28096631
- [Background] Liu-Bryan R, Terkeltaub R. Emerging regulators of the inflammatory process in osteoarthritis. Nat Rev Rheumatol. 2015 Jan;11(1):35-44. doi: 10.1038/nrrheum.2014.162. Epub 2014 Sep 30. PMID 25266449
- [Background] Livshits G, Zhai G, Hart DJ, Kato BS, Wang H, Williams FM, Spector TD. Interleukin-6 is a significant predictor of radiographic knee osteoarthritis: The Chingford Study. Arthritis Rheum. 2009 Jul;60(7):2037-45. doi: 10.1002/art.24598. PMID 19565477
- [Background] Loebel C, Burdick JA. Engineering Stem and Stromal Cell Therapies for Musculoskeletal Tissue Repair. Cell Stem Cell. 2018 Mar 1;22(3):325-339. doi: 10.1016/j.stem.2018.01.014. Epub 2018 Feb 8. PMID 29429944
- [Background] Luyten FP, Vanlauwe J. Tissue engineering approaches for osteoarthritis. Bone. 2012 Aug;51(2):289-96. doi: 10.1016/j.bone.2011.10.007. Epub 2011 Oct 17. PMID 22023933
- [Background] Mabey T, Honsawek S. Cytokines as biochemical markers for knee osteoarthritis. World J Orthop. 2015 Jan 18;6(1):95-105. doi: 10.5312/wjo.v6.i1.95. eCollection 2015 Jan 18. PMID 25621214
- [Background] McCulloch RS, Ashwell MS, Maltecca C, O'Nan AT, Mente PL. Progression of Gene Expression Changes following a Mechanical Injury to Articular Cartilage as a Model of Early Stage Osteoarthritis. Arthritis. 2014;2014:371426. doi: 10.1155/2014/371426. Epub 2014 Nov 16. PMID 25478225
- [Background] Mobasheri A, Matta C, Zakany R, Musumeci G. Chondrosenescence: definition, hallmarks and potential role in the pathogenesis of osteoarthritis. Maturitas. 2015 Mar;80(3):237-44. doi: 10.1016/j.maturitas.2014.12.003. Epub 2014 Dec 24. PMID 25637957
- [Background] Mokbel AN, El Tookhy OS, Shamaa AA, Rashed LA, Sabry D, El Sayed AM. Homing and reparative effect of intra-articular injection of autologus mesenchymal stem cells in osteoarthritic animal model. BMC Musculoskelet Disord. 2011 Nov 15;12:259. doi: 10.1186/1471-2474-12-259. PMID 22085445
- [Background] Montaseri A, Busch F, Mobasheri A, Buhrmann C, Aldinger C, Rad JS, Shakibaei M. IGF-1 and PDGF-bb suppress IL-1beta-induced cartilage degradation through down-regulation of NF-kappaB signaling: involvement of Src/PI-3K/AKT pathway. PLoS One. 2011;6(12):e28663. doi: 10.1371/journal.pone.0028663. Epub 2011 Dec 14. PMID 22194879
- [Background] Moussa M, Lajeunesse D, Hilal G, El Atat O, Haykal G, Serhal R, Chalhoub A, Khalil C, Alaaeddine N. Platelet rich plasma (PRP) induces chondroprotection via increasing autophagy, anti-inflammatory markers, and decreasing apoptosis in human osteoarthritic cartilage. Exp Cell Res. 2017 Mar 1;352(1):146-156. doi: 10.1016/j.yexcr.2017.02.012. Epub 2017 Feb 13. PMID 28202394
- [Background] Murphy JM, Dixon K, Beck S, Fabian D, Feldman A, Barry F. Reduced chondrogenic and adipogenic activity of mesenchymal stem cells from patients with advanced osteoarthritis. Arthritis Rheum. 2002 Mar;46(3):704-13. doi: 10.1002/art.10118. PMID 11920406
- [Background] Murphy JM, Fink DJ, Hunziker EB, Barry FP. Stem cell therapy in a caprine model of osteoarthritis. Arthritis Rheum. 2003 Dec;48(12):3464-74. doi: 10.1002/art.11365. PMID 14673997
- [Background] Osterman C, McCarthy MB, Cote MP, Beitzel K, Bradley J, Polkowski G, Mazzocca AD. Platelet-Rich Plasma Increases Anti-inflammatory Markers in a Human Coculture Model for Osteoarthritis. Am J Sports Med. 2015 Jun;43(6):1474-84. doi: 10.1177/0363546515570463. Epub 2015 Feb 25. PMID 25716226
- [Background] Bum Park Y, Ah Choi W, Kim YK, Chul Lee S, Hae Lee J. Accuracy of blind versus ultrasound-guided suprapatellar bursal injection. J Clin Ultrasound. 2012 Jan;40(1):20-5. doi: 10.1002/jcu.20890. Epub 2011 Oct 28. PMID 22033897
- [Background] Park YB, Ha CW, Kim JA, Han WJ, Rhim JH, Lee HJ, Kim KJ, Park YG, Chung JY. Single-stage cell-based cartilage repair in a rabbit model: cell tracking and in vivo chondrogenesis of human umbilical cord blood-derived mesenchymal stem cells and hyaluronic acid hydrogel composite. Osteoarthritis Cartilage. 2017 Apr;25(4):570-580. doi: 10.1016/j.joca.2016.10.012. Epub 2016 Oct 24. PMID 27789339
- [Background] Patti AM, Gabriele A, Vulcano A, Ramieri MT, Della Rocca C. Effect of hyaluronic acid on human chondrocyte cell lines from articular cartilage. Tissue Cell. 2001 Jun;33(3):294-300. doi: 10.1054/tice.2001.0178. PMID 11469544
- [Background] Purita, Joseph. Lecture Notes in Bio Engineering: Platelet-Rich Plasma. Springer-Verlag Berlin Heidelberg, 2014
- [Background] Quartana PJ, Finan PH, Page GG, Smith MT. Effects of insomnia disorder and knee osteoarthritis on resting and pain-evoked inflammatory markers. Brain Behav Immun. 2015 Jul;47:228-37. doi: 10.1016/j.bbi.2014.12.010. Epub 2014 Dec 20. PMID 25532786
- [Background] Rannou, Francois. Atlas of Osteoarthritis. 2nd ed. London: Springer Healthcare, 2018.
- [Background] Research and Development, Arthrex. "Bone Marrow Aspirate Processing Systems: A Comparison Study." Arthrex Research and Development , 2018.
- [Background] Ruiz M, Maumus M, Fonteneau G, Pers YM, Ferreira R, Dagneaux L, Delfour C, Houard X, Berenbaum F, Rannou F, Jorgensen C, Noel D. TGFbetai is involved in the chondrogenic differentiation of mesenchymal stem cells and is dysregulated in osteoarthritis. Osteoarthritis Cartilage. 2019 Mar;27(3):493-503. doi: 10.1016/j.joca.2018.11.005. Epub 2018 Nov 28. PMID 30502449
- [Background] Sanchez-de-Diego C, Valer JA, Pimenta-Lopes C, Rosa JL, Ventura F. Interplay between BMPs and Reactive Oxygen Species in Cell Signaling and Pathology. Biomolecules. 2019 Sep 26;9(10):534. doi: 10.3390/biom9100534. PMID 31561501
- [Background] Sobacchi C, Palagano E, Villa A, Menale C. Soluble Factors on Stage to Direct Mesenchymal Stem Cells Fate. Front Bioeng Biotechnol. 2017 May 17;5:32. doi: 10.3389/fbioe.2017.00032. eCollection 2017. PMID 28567372
- [Background] Sommerlath K, Lysholm J, Gillquist J. The long-term course after treatment of acute anterior cruciate ligament ruptures. A 9 to 16 year followup. Am J Sports Med. 1991 Mar-Apr;19(2):156-62. doi: 10.1177/036354659101900211. PMID 2039067
- [Background] Southworth TM, Naveen NB, Tauro TM, Leong NL, Cole BJ. The Use of Platelet-Rich Plasma in Symptomatic Knee Osteoarthritis. J Knee Surg. 2019 Jan;32(1):37-45. doi: 10.1055/s-0038-1675170. Epub 2018 Nov 13. PMID 30423591
- [Background] Spees JL, Lee RH, Gregory CA. Mechanisms of mesenchymal stem/stromal cell function. Stem Cell Res Ther. 2016 Aug 31;7(1):125. doi: 10.1186/s13287-016-0363-7. PMID 27581859
- [Background] Srinivasan PP, McCoy SY, Jha AK, Yang W, Jia X, Farach-Carson MC, Kirn-Safran CB. Injectable perlecan domain 1-hyaluronan microgels potentiate the cartilage repair effect of BMP2 in a murine model of early osteoarthritis. Biomed Mater. 2012 Apr;7(2):024109. doi: 10.1088/1748-6041/7/2/024109. Epub 2012 Mar 29. PMID 22455987
- [Background] Sundman EA, Cole BJ, Karas V, Della Valle C, Tetreault MW, Mohammed HO, Fortier LA. The anti-inflammatory and matrix restorative mechanisms of platelet-rich plasma in osteoarthritis. Am J Sports Med. 2014 Jan;42(1):35-41. doi: 10.1177/0363546513507766. Epub 2013 Nov 5. PMID 24192391
- [Background] Tohidnezhad M, Wruck CJ, Slowik A, Kweider N, Beckmann R, Bayer A, Houben A, Brandenburg LO, Varoga D, Sonmez TT, Stoffel M, Jahr H, Lippross S, Pufe T. Role of platelet-released growth factors in detoxification of reactive oxygen species in osteoblasts. Bone. 2014 Aug;65:9-17. doi: 10.1016/j.bone.2014.04.029. Epub 2014 May 4. PMID 24798492
- [Background] Van Pham P, Bui KH, Ngo DQ, Vu NB, Truong NH, Phan NL, Le DM, Duong TD, Nguyen TD, Le VT, Phan NK. Activated platelet-rich plasma improves adipose-derived stem cell transplantation efficiency in injured articular cartilage. Stem Cell Res Ther. 2013 Aug 1;4(4):91. doi: 10.1186/scrt277. PMID 23915433
- [Background] Vangsness CT Jr, Farr J 2nd, Boyd J, Dellaero DT, Mills CR, LeRoux-Williams M. Adult human mesenchymal stem cells delivered via intra-articular injection to the knee following partial medial meniscectomy: a randomized, double-blind, controlled study. J Bone Joint Surg Am. 2014 Jan 15;96(2):90-8. doi: 10.2106/JBJS.M.00058. PMID 24430407
- [Background] Wang Y, Shimmin A, Ghosh P, Marks P, Linklater J, Connell D, Hall S, Skerrett D, Itescu S, Cicuttini FM. Safety, tolerability, clinical, and joint structural outcomes of a single intra-articular injection of allogeneic mesenchymal precursor cells in patients following anterior cruciate ligament reconstruction: a controlled double-blind randomised trial. Arthritis Res Ther. 2017 Aug 2;19(1):180. doi: 10.1186/s13075-017-1391-0. PMID 28768528
- [Background] Wasterlain AS, Braun HJ, Harris AH, Kim HJ, Dragoo JL. The systemic effects of platelet-rich plasma injection. Am J Sports Med. 2013 Jan;41(1):186-93. doi: 10.1177/0363546512466383. Epub 2012 Dec 4. PMID 23211708
- [Background] Webber TA, Webber AE, Matzkin E. Rate of adverse reactions to more than 1 series of viscosupplementation. Orthopedics. 2012 Apr;35(4):e514-9. doi: 10.3928/01477447-20120327-26. PMID 22495852
- [Background] Wu CC, Sheu SY, Hsu LH, Yang KC, Tseng CC, Kuo TF. Intra-articular Injection of platelet-rich fibrin releasates in combination with bone marrow-derived mesenchymal stem cells in the treatment of articular cartilage defects: An in vivo study in rabbits. J Biomed Mater Res B Appl Biomater. 2017 Aug;105(6):1536-1543. doi: 10.1002/jbm.b.33688. Epub 2016 Apr 29. PMID 27125598
- [Background] Wyles CC, Houdek MT, Behfar A, Sierra RJ. Mesenchymal stem cell therapy for osteoarthritis: current perspectives. Stem Cells Cloning. 2015 Aug 28;8:117-24. doi: 10.2147/SCCAA.S68073. eCollection 2015. PMID 26357483